CLINICAL TRIAL: NCT05960565
Title: Glucagon Enhanced Insulin Absorption in Diabetes Mellitus Type 1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: No sign of the anticipated effect.
Sponsor: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EU CT 2022-502455-57-01
Record Dates: First submitted 2023-06-19; First posted 2023-07-25 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Glucagon

STUDY DESIGN:
Intervention Model Description: One day with glucagon and one day without glucagon
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Glucagon (Experimental): Micro dose of glucagon is aded at the insulin injection site
  Interventions: Drug: Glucagon
- Control (No Intervention): Insulin injected without any glucagon

INTERVENTIONS:
Drug: Glucagon — A micro-dose of glucagon is added exactly at the same site as insulin is injected.
  Arms: Glucagon

SUMMARY:
The investigators will study the effect of microdoses of glucagon at the site of subcutaneous insulin injection. The investigators have unpublished data from anesthetized pigs indicating a major enhancement of insulin absorption.

DETAILED DESCRIPTION:
People with type 1 diabetes will come fasting in the morning to the research facility on two separate days. Both days participants will have a breakfast of their own choice and their regular dose of meal insulin injected. Lyumjev will be used. Frequently collected blood sampled will be analysed for glucose, insulin and glucagon for 3.5 hours. The procedures will be exactly the same both days except that on one of the days they will be randomised to a small dose of glucagon that will be injected at exactly the same site as Lyumjev insulin is injected.

ELIGIBILITY:
Inclusion Criteria:

1: Type 1 diabetes for at least 1 year. 2. Age 18 - 70 years. 3. Last known HbA1c <86 mmol/mol. 4. Treated with continuous subcutaneous insulin infusion (CSII) by an insulin pump or multiple daily insulin injections (MDII).

Exclusion Criteria:

1. Pregnant women or women trying to conceive.
2. Any chronic disease, including psychiatric illness, judged incompatible with participation in the study.
3. Unfit for participation for any reason judged by the investigators.
4. Known hypersensitivity to glucagon or any of the excipients of the drug formulation.
5. Known phaeochromocytoma. -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-12-22 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Area under the glucose curve | From time 0 minutes to time 60 minutes
  The area under the glucose curve (change from baseline glucose level)

SECONDARY OUTCOMES:
Area under glucose curve | Any other time span from time 0 minutes to time 180 minutes
  The area under the glucose curve (change from baseline glucose level)
Area under insulin curve | Any time frame from time 0 minutes to time 180 minutes
  The area under the insulin curve
Area under glucagon curve | Any time frame from time 0 minutes to time 180 minutes
  The area under the glucagon curve
Pharmacokinetics of insulin | Start from time 0
  Time to Cmax.
Pharmacokinetics of glucagon | Start from time 0
  Time to Cmax

CONTACTS AND LOCATIONS:
Overall Officials: Sven M Carlsen, MD, PhD, Principal Investigator — St. Olav's University Hospital
Locations (1):
- Department of Endocrinology, St. Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Am MK, Munkerud EY, Berge MH, Christiansen SC, Carlsen SM. The effect of glucagon on local subcutaneous blood flow in non-diabetic volunteers; a proof-of-concept study. Eur J Pharmacol. 2022 Jul 5;926:175045. doi: 10.1016/j.ejphar.2022.175045. Epub 2022 May 21. PMID 35609678
- [Background] Teigen IA, Riaz M, Am MK, Christiansen SC, Carlsen SM. Vasodilatory effects of glucagon: A possible new approach to enhanced subcutaneous insulin absorption in artificial pancreas devices. Front Bioeng Biotechnol. 2022 Sep 21;10:986858. doi: 10.3389/fbioe.2022.986858. eCollection 2022. PMID 36213069